CLINICAL TRIAL: NCT06847841
Title: Cost-Effectiveness and Clinical Outcomes of Double J Stent Versus Percutaneous Feeding Tube Placement Following Open Pyeloplasty in Pediatric Patients: A Prospective Randomized Single-center Study
Acronym: DJS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hayat Abad Medical Complex, Peshawar (Other Government)
Responsible Party: Principal Investigator, Abdul Haseeb, Post graduate resident, Hayat Abad Medical Complex, Peshawar
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2376/HMC-QAD-F; Institute of Kidney Diseases (Other: Institute of Kidney Diseases, Hayatabad Medical Complex)
Record Dates: First submitted 2025-02-21; First posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Pyeloplasty; Complications of Surgical Procedures or Medical Care; Hospital Stay
Keywords: Pyleoplasty; Hospital Stay; Complications; DJS; PUJO

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PUJO (Active Comparator): Patients having PUJ Obstruction and booked for open pyeloplasty
  Interventions: Procedure: Double J Stent Placement; Procedure: Percutaneous Feeding Tube Placement

INTERVENTIONS:
Procedure: Double J Stent Placement — Patient in whom a DJS will be placed for post op drainage
Procedure: Percutaneous Feeding Tube Placement — Patient in whom a PrcFT will be placed for post op drainage

SUMMARY:
Open pyeloplasty is a common surgical intervention for pediatric patients with ureteropelvic junction obstruction. Post-operative management strategies, including the use of a double J stent and a percutaneous feeding tube, vary widely. While both options have demonstrated effectiveness in drainage, their relative clinical outcomes, costs, and overall value in pediatric urology remain unclear. This randomized controlled trial (RCT) aims to compare the clinical efficacy and cost-effectiveness of these two post-operative interventions in pediatric patients undergoing open pyeloplasty.

DETAILED DESCRIPTION:
This is going to be a prospective randomized study of pediatric patients undergoing open pyeloplasty in Department of Pediatric Urology, Institute of Kidney Diseases, Peshawar. After obtaining approval from the ethical committee board of the hospital. The aim and benefits of the study will be well explained to the parents of all the patients, and they will be briefed as well that no risk is involved while participating in this study. Then informed consent will be obtained and the patients will be randomly assigned to receive either a double J stent or a percutaneous feeding tube for post-operative drainage. Randomization will be performed using block randomization to ensure balance between groups. A mix of both consecutive and purposive sampling technique to recruit patient until the desire sample size is reached. The primary outcomes included pain relief, the rate of complications like post op infection, obstruction, and length of hospital stay. Secondary outcomes included incidence of re-operations, and cost analysis of the two interventions. A cost-effectiveness analysis will be conducted from the healthcare provider's perspective, considering direct medical costs (surgical, hospitalization, and follow-up care) and the quality-adjusted life years (QALYs) for each group. Data will be analyses using SPSS and results will be reported

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary PUJO and outflow obstruction on renal Scan who are candidates for elective open pyeloplasty

Exclusion Criteria:

* Patients who are previous operated for PUJO , and having recurrence

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2025-07-10 (Estimated); Study Completion 2025-07-10 (Estimated)

PRIMARY OUTCOMES:
Complication Rate | up to 4 weeks on post follow up on clinical examination and relevant investigations
  Rate of Complication including pain, bleeding, re operation

SECONDARY OUTCOMES:
Cost Effectiveness | one month on post follow up on clinical examination and relevant investigation
  Whether PrcFT is cost effective than DJS or not

CONTACTS AND LOCATIONS:
Overall Officials: Abdul Haseeb, MBBS, MRCS, Principal Investigator — Institute Of kidney Diseases
Locations (1):
- Institute of Kidney Disease., Peshawar, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
As part of our commitment to research transparency and data-sharing practices, we plan to share individual participant data (IPD) obtained from this clinical trial. The purpose of sharing IPD is to enable further research, facilitate meta-analyses, and contribute to scientific advancements that can improve patient care and clinical outcomes. Scope of Data to be Shared
  The de-identified individual participant data that will be shared includes:
  Demographic details such as age, sex, and relevant baseline characteristics Clinical and laboratory data collected during the study Outcome measures related to the study objectives Adverse event reports and safety data All shared data will be de-identified to ensure participant confidentiality and privacy in accordance with applicable ethical guidelines and regulatory requirements.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: The data will be made publicly available six months after the primary study results are published in a peer-reviewed journal. The dataset will remain accessible for a period of five years from the initial release, after which continued access will be evaluated based on scientific interest and data usage
Access Criteria: The IPD will be stored in a secure, electronic form with the principal investigator.
  Researchers interested in accessing the data will be required to submit a request to the principal author via this email: ahaseeb.dr@gmail.com Conditions for Data Access Access to the shared data will be granted to qualified researchers affiliated with recognized academic or clinical institutions. Interested researchers must submit a methodologically sound research proposal outlining the objectives and intended use of the data. Approval will be based on scientific merit and alignment with ethical standards.
  Before access is granted, researchers will be required to:
  Sign a Data Use Agreement (DUA) to ensure appropriate use of the dataset Agree to maintain confidentiality and not attempt to re-identify participants Provide a commitment to acknowledge the original study and funding sources in any resulting publications